CLINICAL TRIAL: NCT07042815
Title: Multi Site Long-term Follow-up for Those With Experimental Epidural Stimulation After Severe Spinal Cord Injury
Brief Title: Long-term Follow-up for Epidural Stimulation in SCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Gail Forrest, Director, Tim and Caroline Reynolds Center for Spinal Stimulation, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R-1273-24
Record Dates: First submitted 2025-04-28; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: SCI - Spinal Cord Injury
Keywords: spinal stimulation; epidural
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participants will receive the same stimulation programs and assessments as they did during the previous study they were enrolled in. This model is tracking the participant longitudinally at di intervals of 6 months and 1 year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Home Use and Follow-Up Visit Group (Experimental): Participants will be cleared by study staff for home-use of the stimulation programs they received in the previous study. Participants will then follow and log the programs according to study staff recommendations.
  Interventions: Device: Epidural Stimulation Programs

INTERVENTIONS:
Device: Epidural Stimulation Programs — Epidural stimulations will accompany stimulation programs that have been established during research visits in the prior study and have been recommended by the clinical research team for use in the home and community. Stimulation programs will be given for activities (such as standing or walking) and/or responses that were completed in the previous study. This will be continued until the device is removed or approved for commercial use.

SUMMARY:
The goal of this study is to understand long-term effects of spinal cord stimulation in individuals who have a spinal cord injury. The main aims are to:

1. provide support for those with epidural stimulators who choose to continue stimulating because they deemed them to improve their quality of life
2. provide additional sites for follow-up so that the financial burden can be minimized for the research participants to travel
3. collect long-term safety data; and
4. when feasible collect data to understand the sustainability of outcomes.

Participants will:

* receive stimulation programs and software for the activities and/or functions completed in the previous study and demonstrate to the research staff that I can conduct them without their help to use at home
* continue using the stimulation programs at home as directed by the research staff
* return to Kessler Foundation for a follow-up visit (approx. 2 hours) with assessments at 6 months, 1 year, and once a year after enrolled in the follow-up study last until either the device is turned off, removed or the device is commercially approved.

DETAILED DESCRIPTION:
SCI participants who previously had an epidural stimulation device and completed the initial study can continue using stimulation programs at home once they have proven to study staff that they can use the programs and device on their own. This follow-up study will give insight into potential benefits from long-term use of spinal stimulation.

In-person follow-up visits (approx. 2 hours long) will be requested at 6-months, 1 year, and once a year until the device is removed or approved for commercial use. If the participant can't come to Kessler for an in-person visit, a remote tele-health visit will be arranged. Visits include:

* medical history since the last visit will be collected
* a physical exam
* assessments completed during the study previously enrolled in including:

  * Testing of muscle and limb responses to stimulation
  * Assessment of sitting, standing, and stepping function
  * Bladder and bowel function tests
  * Spasticity assessments
  * Blood pressure monitoring
  * Questionnaires
  * MRI
  * TMS
  * DXA
* The study physician will contribute to decisions about which of these assessments are most appropriate to perform at a particular visit
* The investigators will review stimulation logs
* The investigator will review results of the assessments and discuss continuing in the follow up study.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* have a spinal cord injury that is not getting worse
* received a neurostimulator and electrode array as part of a previous study
* choose to continue epidural stimulation in the home and community
* have completed a previous IRB approved epidural stimulation study at a participating research site

Exclusion Criteria:

* heart, lung, bladder, kidney or other untreated medical disorder unrelated to SCI
* choose not to use the epidural stimulation as recommended by the investigators
* withdrawn from the main epidural stimulation study or made the choice to remove the stimulator/return the controller to the site
* new surgeries, diagnoses, or other changes in status since completion of main epidural study that may affect the ability to complete assessments
* Unable to undergo an MRI
* Conditions that may make me ineligible for transcranial magnetic stimulation (a kind of brain stimulation through the skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Motor Control Assessments with stimulation | On average, 1 hour each visit completed 6 months, 1 year, and yearly
  Participants will receive epidural stimulation and motor tasks based on their prior study participations' assessments and programming. During this stimulation, participants will be given motor tasks that may involve sitting, standing, stepping, and movement of their extremities. Electrodes will be placed over the specific muscles measured in that motor task. Data from those electrode readings will be transferred to numerical data. Plots from that numerical data will be created by identifying amplitude against stimulation intensity and threshold intensity, rate of recruitment, and plateau intensity per muscle using customized MATLAB software and then compared to results in the participants' prior training study.
Bladder Function Assessment | on average, 30 minutes each visit completed 6 months, 1 year, and yearly
  This assessment will only be performed in the participants who previously completed the locomotor, bladder and bowel intervention study (R-1230-23) The bladder function assessment includes a urinalysis and bladder pressure test. The bladder pressure test involves emptying of the bladder and refilling with saline with a catheter that measures bladder pressure. Urinalysis is to screen for bacteria. Results will be recorded and compared with previous study data.
Cardiovascular Assessment | 24 hours prior to visit, completed 6 months, 1 year, and yearly
  Participant blood pressure will be monitored over a 24-hour period outside the lab with a blood pressure monitor provided by the lab and during visit assessments. The reading will be recorded and compared to prior study readings.

SECONDARY OUTCOMES:
Questionnaires | On average, 30 minutes each visit completed 6 months, 1 year, and yearly
  All participants, regardless of prior training group will complete a series of questionnaires about their overall functioning at each follow-up visit. The questionnaires cover general topics about quality of life including perceived quality of life, experiences using the home stimulation program, and sexual (male or female), bladder and bowel function. These are multiple choice questions, with each answer valued between 0 and 5 points for all except the quality of life section, where answer scores vary based on question and has an overall score of 0-100.
  An aggregate score for each domain will be compiled and compared with recorded scores from before, during, and directly after the training portion of the study they previously completed as a secondary measure of comparison to the assessment results.
Imaging Assessments | On Average, 15 minutes each visit completed 6 months, 1 year, and yearly
  Participants may be asked to repeat imaging assessments that were performed during their previous intervention study such as a Dual-energy X-ray absorptiometry (DXA) and/or MRI. Imaging data will be compared to prior imaging to monitor for any changes.
Spasticity Monitoring | Each visit completed 6 months, 1 year, and yearly
  Each participant is assigned an observer to accompany the research participant on their visits. The responsibility of the observer is to communicate with the research participant and monitor their well-being. The observer, the technicians, the research nurse and/or the research physical therapist will monitor the research participant at each visit for spasticity events. If a participant experiences a spasticity event during any training, a member of the study team will visually monitor the spasm and record the duration, location, and level of pain the participant is experiencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data